CLINICAL TRIAL: NCT00695981
Title: The Effectiveness and Cost-Effectiveness of Operative and Non-operative Management of Rotator Cuff Tear
Brief Title: Operative Versus Non-operative Management of Rotator Cuff Tear
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: Academy of Finland (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Juha Paloneva, Md, PhD, Central Finland Hospital District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B07103-2
Record Dates: First submitted 2008-03-17; First posted 2008-06-12 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff; Arthroscopic surgery; Open surgery; Physiotherapy; Physical therapy; Effectiveness; RCT; cost-effectiveness
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Conservative Treatment; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotator cuff repair (Active Comparator): Surgery following a 3 months period of active non-operative treatment
  Interventions: Procedure: Rotator cuff repair
- Conservative treatment (Active Comparator): Physiotherapy according to a standardized protocol following a 3 months period of active non-operative treatment
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Rotator cuff repair — Rotator cuff repair + physical therapy according to a standardized protocol
  Other Names: Arthroscopic or open rotator cuff repair
  Arms: Rotator cuff repair
Procedure: Conservative treatment — Physiotherapy according to a standardized protocol
  Other Names: Physical therapy; Non-operative treatment
  Arms: Conservative treatment

SUMMARY:
This study aims at determining the effectiveness and cost-effectiveness of surgical management of full-thickness rotator cuff tears compared to conservative treatment. The research setting is prospective, randomised, and controlled.

The aim of the study is to search out evidence based data of indications for rotator cuff repair. The investigators also aim at offering patients the most efficient and effective treatment and reduce the number of operations that do not have sufficient effectiveness. The data obtained will facilitate developing guidelines for referrals to a specialist when rotator cuff tear is suspected.

The investigators hypothesize that there are subgroups of patients suffering from rotator cuff tears that benefit from surgery whereas other subgroups are best treated conservatively.

DETAILED DESCRIPTION:
Subgroup analyses:

* age
* sex
* duration of symptoms
* presence of trauma before symptoms
* size of tear
* degenerative findings
* other findings in MRI or arthroscopy
* type of operation
* co-morbidities
* occupation
* pain (VAS)
* objective shoulder function
* activities of daily living

ELIGIBILITY:
Inclusion Criteria:

* age over 35 years old
* duration of symptoms at least three months despite of non-operative treatment
* the patient accepts both treatment options (operative and conservative)
* a full-thickness rotator cuff tear in MRI arthrography

Exclusion Criteria:

* previous shoulder operations
* too high risk for operation
* any disease or social problem reducing the ability to co-operate
* rheumatoid arthritis
* severe arthrosis of the glenohumeral or acromioclavicular joint
* irreparable rotator cuff tear (including rotator cuff tear arthropathy)
* progressive malign disease
* adhesive capsulitis
* high-energy trauma before symptoms
* cervical syndrome
* shoulder instability

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain (VAS) and objective shoulder function (Constant score) | 24 months
  VAS (0 to 100 mm), Constant score (0 to 100 points)

SECONDARY OUTCOMES:
Change in pain (VAS) and objective shoulder function (Constant score) | 3 months
  VAS (0 to 100 mm), Constant score (0 to 100 points)
Change in pain (VAS) and objective shoulder function (Constant score) | 6 months
  VAS (0 to 100 mm), Constant score (0 to 100 points)
Change in pain (VAS) and objective shoulder function (Constant score) | 12 months
  VAS (0 to 100 mm), Constant score (0 to 100 points)
Change in pain (VAS) and objective shoulder function (Constant score) | 5 years
  VAS (0 to 100 mm), Constant score (0 to 100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Juha Paloneva, MD, PhD, Principal Investigator — Central Finland Health Care District, University of Eastern Finland
Locations (3):
- Finland (3):
  - University of Helsinki, Helsinki
  - Central Finland Hospital, Jyväskylä
  - Oulu University Hospital, Oulu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oh LS, Wolf BR, Hall MP, Levy BA, Marx RG. Indications for rotator cuff repair: a systematic review. Clin Orthop Relat Res. 2007 Feb;455:52-63. doi: 10.1097/BLO.0b013e31802fc175. PMID 17179786
- [Background] Kukkonen J, Joukainen A, Lehtinen J, Mattila KT, Tuominen EK, Kauko T, Aarimaa V. Treatment of Nontraumatic Rotator Cuff Tears: A Randomized Controlled Trial with Two Years of Clinical and Imaging Follow-up. J Bone Joint Surg Am. 2015 Nov 4;97(21):1729-37. doi: 10.2106/JBJS.N.01051. PMID 26537160
- [Background] Kukkonen J, Joukainen A, Lehtinen J, Mattila KT, Tuominen EK, Kauko T, Aarimaa V. Treatment of non-traumatic rotator cuff tears: A randomised controlled trial with one-year clinical results. Bone Joint J. 2014 Jan;96-B(1):75-81. doi: 10.1302/0301-620X.96B1.32168. PMID 24395315
- [Background] Lambers Heerspink FO, van Raay JJ, Koorevaar RC, van Eerden PJ, Westerbeek RE, van 't Riet E, van den Akker-Scheek I, Diercks RL. Comparing surgical repair with conservative treatment for degenerative rotator cuff tears: a randomized controlled trial. J Shoulder Elbow Surg. 2015 Aug;24(8):1274-81. doi: 10.1016/j.jse.2015.05.040. PMID 26189808
- [Background] Moosmayer S, Lund G, Seljom US, Haldorsen B, Svege IC, Hennig T, Pripp AH, Smith HJ. Tendon repair compared with physiotherapy in the treatment of rotator cuff tears: a randomized controlled study in 103 cases with a five-year follow-up. J Bone Joint Surg Am. 2014 Sep 17;96(18):1504-14. doi: 10.2106/JBJS.M.01393. PMID 25232074
- [Background] Moosmayer S, Lund G, Seljom U, Svege I, Hennig T, Tariq R, Smith HJ. Comparison between surgery and physiotherapy in the treatment of small and medium-sized tears of the rotator cuff: A randomised controlled study of 103 patients with one-year follow-up. J Bone Joint Surg Br. 2010 Jan;92(1):83-91. doi: 10.1302/0301-620X.92B1.22609. PMID 20044684
- [Background] Paloneva J, Lepola V, Aarimaa V, Joukainen A, Ylinen J, Mattila VM. Increasing incidence of rotator cuff repairs--A nationwide registry study in Finland. BMC Musculoskelet Disord. 2015 Aug 12;16:189. doi: 10.1186/s12891-015-0639-6. PMID 26265152
- [Background] Paloneva J, Lepola V, Karppinen J, Ylinen J, Aarimaa V, Mattila VM. Declining incidence of acromioplasty in Finland. Acta Orthop. 2015 Apr;86(2):220-4. doi: 10.3109/17453674.2014.977703. Epub 2014 Oct 23. PMID 25340548
- [Derived] Cederqvist S, Flinkkila T, Sormaala M, Ylinen J, Kautiainen H, Irmola T, Lehtokangas H, Liukkonen J, Pamilo K, Ridanpaa T, Sirnio K, Leppilahti J, Kiviranta I, Paloneva J. Non-surgical and surgical treatments for rotator cuff disease: a pragmatic randomised clinical trial with 2-year follow-up after initial rehabilitation. Ann Rheum Dis. 2021 Jun;80(6):796-802. doi: 10.1136/annrheumdis-2020-219099. Epub 2020 Dec 3. PMID 33272959
- See also: Clinical Musculoskeletal Diseases Research Group internet pages — http://www.ksshp.fi/musculoskeletalresearch